CLINICAL TRIAL: NCT03121950
Title: Movement and Music Intervention for Individuals With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Deb Kegelmeyer, Professor Clinical, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016H0211
Record Dates: First submitted 2017-04-10; First posted 2017-04-20 (Actual); Results first posted 2019-06-20 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Dementia With Lewy Bodies; Dementia
Keywords: dementia
MeSH Terms: conditions — Lewy Body Disease; Dementia | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be placed in one of two groups. One group will participate 2 times a week in a dance class. The other group will listen to live music once a week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance in dementia (Experimental): examine if participating in a dance class improves mobility and/or cognition in individuals with dementia.
  Interventions: Other: Dance
- Music and dementia (Active Comparator): examine if listening to music improves mobility and/or cognition in individuals with dementia.
  Interventions: Other: Music

INTERVENTIONS:
Other: Dance — The primary intervention is a dance class
  Arms: Dance in dementia
Other: Music — the secondary intervention is listening to live music
  Arms: Music and dementia

SUMMARY:
The goal of the study is to learn about how possible benefits of movement and music for individuals with dementia. Individuals with dementia will participate in a dance class. The study includes assessments of walking, balance and cognition.

DETAILED DESCRIPTION:
Dementia impacts 5%-7% of individuals >60 years old. It impacts the person's ability to perform work, care for him/herself and ultimately leads to physical disability. There is a high caregiver burden associated with dementia and many individuals require care in a long-term care facility. There is some emerging evidence that music based interventions may have a protective effect on the brain in those with dementia. There is also evidence that doing activities that engage the brain through music are beneficial. This study seeks to investigate the potential benefits of a music based intervention for individuals with dementia. The study aims to recruit individuals with a diagnosis of dementia. Once enrolled participants will undergo assessment of walking, balance and cognition and then be asked to participate either in a dance class or to listen to live music. After 6 weeks and again at the end of the study (after 12 weeks) participants will undergo assessments of walking, balance and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia
* Mini-Mental State Examination score > 9
* Age > 60 years
* Able to follow simple instructions

Exclusion Criteria:

* Unable to walk 10 feet unassisted
* Presence of orthopedic disorder that impacts walking
* Presence of other neurologic diagnosis that impacts cognitive or motor function such as stroke, Parkinson disease or traumatic brain injury

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deb Kegelmeyer, DPT, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was excluded due to not meeting criteria on minimum score required for participation on the Mini Mental Status Examination
Period: Overall Study
Arm/Group | Dance in Dementia | Music and Dementia
Started | 17 | 3
Completed | 6 | 1
Not Completed | 11 | 2
Not completed — Withdrawal by Subject | 11 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dance in Dementia | Music and Dementia | Total
Number analyzed (Participants) | 17 | 3 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 17 | 3 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.76 (7.55) | 74 (11.36) | 82.3 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 8 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 3 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Timed up and go Cognitive
Description: The change in time to complete the Timed Up and Go - Cognitive (TUG-Cog) is recorded in seconds. The participant is timed with a stop watch while walking 3 meters turning and returning to a chair while performing a concurrent cognitive task. This time is compared to the Timed Up and Go (TUG) and the difference in time indicates the effect cognitive deficits have on motor function. Higher scores, indicating more time, means worse outcomes.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dance in Dementia | Music and Dementia
Number analyzed (Participants) | 6 | 1
seconds | -6.49 (9.66) | -13.35 (0)

2. Secondary Outcome: Change in Score on the Montreal Cognitive Assessment
Description: The Montreal Cognitive Assessment (MoCA) is an assessment of overall cognitive status. The range of scores is 0-30, with higher scores indicating better outcomes. Scores 26 or higher indicates normal cognitive function.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance in Dementia | Music and Dementia
Number analyzed (Participants) | 6 | 1
score on a scale | -1.5 (2.07) | 0 (0)

3. Other Pre Specified Outcome: Change in Score on the Caregiver Burden Scale
Description: A questionnaire asking caregivers about the impact of caregiving on daily life. Scores range from 0-88, with higher scores indicating worse outcomes or more burden. Scores of 0-20 = little or no burden, 21-40 = mild to moderate burden, 41-60 = moderate to severe burden, and 61-80 = severe burden.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance in Dementia | Music and Dementia
Number analyzed (Participants) | 6 | 1
score on a scale | -5.17 (8.51) | -7 (0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dance in Dementia | Music and Dementia
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/3
Other Adverse Events (participants affected / at risk) | 0/17 | 0/3

LIMITATIONS AND CAVEATS:
Our study had many limitations including significant barriers to recruitment and retention of participants. Because of this, we changed the design to a pretest-posttest pilot study and included data from a participant at 6 weeks in the manuscript.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT03121950/Prot_SAP_ICF_001.pdf